CLINICAL TRIAL: NCT04451057
Title: High Flow Nasal Cannula in Pediatric Patients After Cardiothoracic Surgery:A Randomized Controlled Trial
Brief Title: High Flow Nasal Cannula in Pediatric Patients After Cardiothoracic Surgery
Acronym: OSACA CATS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Osaka University (Other)
Collaborators: Osaka Women's and Children's Hospital (Unknown); Hyogo Prefectural Kobe Children's Hospital (Other); Osaka City General Hospital (Other); Aichi Children's Health and Medical Center (Unknown); National Center for Child Health and Development (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OSACA CATS
Record Dates: First submitted 2020-06-21; First posted 2020-06-30 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-02

CONDITIONS: Pediatric Patients After Cardiothoracic Surgery
Keywords: high flow nasal cannula; conventional oxygen therapy; treatment failure after extubation

STUDY DESIGN:
Intervention Model Description: control group:conventional oxygen therapy interventional group:high flow nasal cannula
Who Masked: Participant
Masking Description: Single blind .Participants and their legal representatives are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high flow nasal nasal cannula (Experimental): Patients allocated for this arm are received high flow nasal cannula therapy after extubation.
  Interventions: Device: high flow nasal cannula therapy
- low flow nasal cannula (Active Comparator): Patients allocated for this arm are received conventional oxygen therapy after extubation.
  Interventions: Device: low flow nasal cannula therapy

INTERVENTIONS:
Device: high flow nasal cannula therapy — Once extubation has taken place, the child will be placed either on conventional oxygen therapy or high flow nasal cannulae according to randomization
  Other Names: high flow nasal cannula oxygen therapy
  Arms: high flow nasal nasal cannula
Device: low flow nasal cannula therapy — Once extubation has taken place, the child will be placed either on conventional oxygen therapy or high flow nasal cannulae according to randomization
  Other Names: conventional oxygen therapy
  Arms: low flow nasal cannula

SUMMARY:
High flow nasal cannula(HFNC) ventilation can provide such effects as wash-out effect of the carbon dioxide inside the anatomical dead space,some level of continuous airway pressure and humidified oxygen gases.

Therefore because of its physiological benefits, it has been reported that HFNC can reduce "treatment failure" after extubation in pediatric patients like preterm babies,or infants who suffer from bronchitis.

However there is no evidence showing that HFNC can reduce "treatment failure" after extubation in pediatric patients after cardiothoracic surgery.

This multi-center randomized controlled trial (RCT) involving pediatric patients after cardiothoracic surgery will be conducted to determine whether HFNC,compared with conventional oxygen therapy,after extubation can reduce the rate of"escalation of care due to treatment failure".

DETAILED DESCRIPTION:
The multi-center RCT will enroll 380 pediatric patients after cardiothoracic surgery from the Intensive Care Units (ICUs) in Japan.Informed consent will be obtained from the their parents or legally representatives.They will receive postoperative standard care in ICU and spontaneous breathing test(SBT).If SBT will be done successfully,they will be extubated.Just before extubation,they will be divided randomly into the intervention group or the control group.After randomization,they will be extubated.After extubation,the intervention group will receive HFNC therapy,while the control group will receive conventional oxygen therapy.The flow in the intervention group will surely be maintained to be high,while the flow in control group will surely be less than 2 liter/min.In both groups,outcome measure will be assessed within 72 hours after extubation,or during ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients younger than two years old after cardiothoracic surgery
* pediatric patients who have been ventilated for more than 12 hours after surgery

Exclusion Criteria:

* patients with tracheostomy
* patients with do-not-resuscitate (DNR)
* patients who have be treated by noninvasive positive pressure ventilation or high flow nasal cannula before surgery
* patients who undergo unplanned extubation
* patients who have withdrawn consent from their legal guardian
* patients who don't need oxygen therapy
* patients who are planned to receive treatment with noninvasive positive pressure ventilation after extubation
* patients who are planned to inhale nitric oxide(NO) after extubation

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 286 (Estimated)
Dates: Start 2020-08-11 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
the rate of"escalation of care due to treatment failure" within 72 hours after extubation | Final outcome measure is assessed when total patients have been recruited.Outcome measure is assessed within 72 hours after extubation.

SECONDARY OUTCOMES:
non event rate within 72 hours after extubation | Final outcome measure is assessed when total patients have been recruited.Outcome measure is assessed within 72 hours after extubation.
  The event is defined as "escalation of care due to treatment failure "after extubation.Non event is defined as other than this event.
peripheral oxygen saturation | Final outcome measure is assessed when total patients have been recruited.Outcome measure is assessed before extubation,1 hour,12 hours,24 hours,48 hours and 72 hours after extubation.
  oxygen saturation (SpO2)
arterial blood gas | Final outcome measure is assessed when total patients have been recruited.Outcome measure is assessed before extubation,1 hour,12 hours,24 hours,48 hours and 72 hours after extubation.
  potential of hydrogen (pH)
arterial blood gas | Final outcome measure is assessed when patients have been recruited.Outcome measure is assessed before extubation,1 hour,12 hours,24 hours,48 hours and 72 hours after extubation.
  partial pressure of carbon dioxide in arterial blood(PaCO2)
arterial blood gas | Final outcome measure is assessed when total patients have been recruited.Outcome measure is assessed before extubation,1 hour,12 hours,24 hours,48 hours and 72 hours after extubation.
  lactate
vital sign | Final outcome measure is assessed when total patients have been recruited.Outcome measure is assessed before extubation,1 hour,12 hours,24 hours,48 hours and 72 hours after extubation.
  respiratory rate
vital sign | Final outcome measure is assessed when total patients have been recruited.Outcome measure is assessed before extubation,1 hour,12 hours,24 hours,48 hours and 72 hours after extubation.
  heart rate
vital sign | Final outcome measure is assessed when total patients have been recruited.Outcome measure is assessed before extubation,1 hour,12 hours,24 hours,48 hours and 72 hours after extubation.
  mean blood pressure
fractional inspired oxygen | Final outcome measure is assessed when total patients have been recruited.Outcome measure is assessed before extubation,1 hour,12 hours,24 hours,48 hours and 72 hours after extubation.
  fractional inspired oxygen (FiO2)
Catecholamine score | Final outcome measure is assessed when total patients have been recruited.Outcome measure is assessed before extubation,1 hour,12 hours,24 hours,48 hours and 72 hours after extubation.
sedative dose | Outcome is assessed like as follows;total dose from 6 hours before extubation to extubation,total dose from 18 hours to 24 hours after extubation,total dose from 42 hours to 48 hours after extubation,total dose from 66 hours to 72 hours after extubation.
Chest x-ray score | Outcome is assessed within 24 hours before extubation,within 24 hours after extubation.
  The presence of atelectasis is expressed by a 5 point score:clear lung fields 0,plate-like atelectasis or slight infiltration 1,partial atelectasis 2,lobar atelectasis 3,bilateral lobar atelectasis 4.
Oxygen flow rate | Outcome is assessed at the time as follows;1 hour,12 hours,24 hours,48 hours and 72 hours after extubation.
  Inhaled oxygen flow rate
criteria of "treatment failure" | Outcome measure is assessed within 72 hours after extubation.
  This criteria of "treatment failure" is defined as follows; 1 tachypnea,2 hypercapnia,3 reduced oxygen saturation,4 tachycardia,5 clinical symptoms suggesting respiratory distress, 6 life threatening signs,7 other clinical concerns or reasons.
Details of"escalation of care" | Outcome measure is assessed within 72 hours after extubation.
  The details of "escalation of care" are defined as follows;"escalation of care" is defined as noninvasive positive pressure ventilation (NPPV) therapy or mechanical ventilation therapy ,if patients have been allocated to intervention group ( group for HFNC therapy ).On the other hand, " escalation of care" is defined as HFNC therapy,NPPV therapy,or mechanical ventilation therapy, if patients have been allocated to control group ( group for conventional oxygen therapy).
at the time of 72 hours after extubation, treatment outcome of the patients who have been diagnosed as "treatment failure" | Outcome measure is assessed at the time of 72 hours after extubation
  This treatment outcome of these patients is defined as follows;1 They haven't receive more"escalation of care" by receiving HFNC therapy,2 They have received noninvasive positive pressure ventilation (NPPV) therapy despite receiving HFNC therapy,3 They have received mechanical ventilation therapy despite receiving HFNC therapy,4They haven't receive more"escalation of care" by receiving NPPV therapy,5 They have received mechanical ventilation therapy despite receiving NPPV therapy.
the rate of reintubation at the time of 72 hours after extubation | Outcome measure is assessed at the time of 72 hours after extubation
the length of ICU stay | through study completion,an average of 1 month
the length of hospital stay | Outcome measure is assessed when the patients is discharged from the hospital or the time of six months after extubation.
adverse events | through study completion,an average of 1 month
prespecified sub group analysis | Final outcome measure is assessed when total patients have been recruited.Outcome measure is assessed within 72 hours after extubation.
  Primary outcome is assessed by sub group analysis as follows; age(less than 30 days,more than 31 days).
prespecified sub group analysis | Final outcome measure is assessed when total patients have been recruited.Outcome measure is assessed within 72 hours after extubation.
  Primary outcome is assessed by sub group analysis as follows;chromosomal abnormality.
prespecified sub group analysis | Final outcome measure is assessed when total patients have been recruited.Outcome measure is assessed within 72 hours after extubation.
  Primary outcome is assessed by sub group analysis as follows;RACHES-1 score. hours,more than 6 hours)
prespecified sub group analysis | Final outcome measure is assessed when total patients have been recruited.Outcome measure is assessed within 72 hours after extubation.
  Primary outcome is assessed by sub group analysis as follows;postoperative cyanosis.
prespecified sub group analysis | Final outcome measure is assessed when total patients have been recruited.Outcome measure is assessed within 72 hours after extubation.
  Primary outcome is assessed by sub group analysis as follows; operation time(less than 6 hours,more than 6 hours).

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Yoshida, MDPhD, Study Chair — Department of Anesthesiology and Intensive Care Medicine, Osaka University
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, Osaka University, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No